CLINICAL TRIAL: NCT04508374
Title: Intralesional Diode Laser Treatment of Fistulas in Hidradenitis Suppurativa: Protocol for a Within-person Randomised Trial
Brief Title: Intralesional Diode Laser Treatment of Fistulas in Hidradenitis Suppurativa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Gregor Jemec, Professor, PhD, DmsC, Head of Dpt., Zealand University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 19- 001165
Record Dates: First submitted 2020-08-02; First posted 2020-08-11 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Intervention Model Description: The study is designed as a randomised, contralaterally-controlled, within-person design, where HS patients are randomised to undergo intralesional laser fibre treatment of HS tunnels in either right or left side of the body, whereas the other tunnel is left as an untreated control.
Who Masked: Outcomes Assessor
Masking Description: Evaluation of clinical photos and percentage closure by Ultrasound will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1470 nm diode laser treatment of right HS-fistula (Experimental): This is an intra-person study, comparing outcomes within participants. All participants will receive active 1470 nm intra-lesional diode laser treatment on one HS tunnel. Half of the enroled patients will receive active treatment of the right side, while the HS tunnel on the left side will be left as an untreated control.
  Interventions: Procedure: 1470 nm intra-lesional diode laser treatment of right HS tunnel
- 1470 nm diode laser treatment of left HS-fistula (Experimental): This is an intra-person study, comparing outcomes within participants. All participants will receive active 1470 nm intra-lesional diode laser treatment on one HS tunnel. Half of the enroled patients will receive active treatment of the left side, while the HS tunnel on the right side will be left as an untreated control.
  Interventions: Procedure: 1470 nm intra-lesional diode laser treatment of left HS tunnel

INTERVENTIONS:
Procedure: 1470 nm intra-lesional diode laser treatment of right HS tunnel — Ten patients: 1470 nm intra-lesional diode laser treatment of right HS-tunnel randomized to active treatment.
  Arms: 1470 nm diode laser treatment of right HS-fistula
Procedure: 1470 nm intra-lesional diode laser treatment of left HS tunnel — Ten patients: 1470 nm intra-lesional diode laser treatment of left HS-tunnel randomized to active treatment.
  Arms: 1470 nm diode laser treatment of left HS-fistula

SUMMARY:
Hidradenitis suppurativa (HS) is a common chronic skin disease where patients experience inflamed painful nodules and chronic suppurating tunnels under the skin that often leave mutilating scars. Symptoms typically begin during adolescence and patients struggle with pain, pruritus, malodor and purulent discharge compromising work life, physical exercise, and sexual habits. Consequently, the risk of social exclusion, anxiety, depression, and suicide is increased among patients suffering from HS.

Creams, tablets, and injections aim to gain disease control, yet are sometimes not sufficient. Once HS tunnels have formed, surgical intervention is often required.

Recently, emergence of flexible diode laser fibers has enabled treatment of tunnels from within. The technique has been tested for perianal tunnels and in few studies also for HS tunnels with promising results. Overall, the laser fiber technique is still new, and knowledge of optimal treatment settings is sparse. However, there is reason to believe that intralesional laser fiber treatment of HS tunnels may provide a new tissue-sparing alternative to conventional surgical techniques with a potential to produce fewer side effects, less scaring, shorter downtime after surgery and possibly, also improved inflammatory control.

This study aims to investigate the efficacy and safety of laser fiber treatment of HS tunnels.

Method The project is carried out at the Dermatological Department, Roskilde University Hospital under the leadership of principal investigator Professor DmSc Gregor Jemec.

A prospective cohort study of intralesional laser fiber treatment of HS fistulas is planned.

After signing informed consent, patients with two comparable HS tunnels in typical areas will draw lot to receive experimental laser fiber treatment of one tunnel while the other tunnel serve as control. Efficacy will be monitored by pain scores, ultrasound, clinical photos, clinical measures of disease activity, quality-of-life scores, and skin biopsies. Patients will be followed 2, 6, 12 weeks and if possible, also 52 weeks after treatment. After 12 weeks, patients will be offered laser fiber treatment or standard of care surgery to the untreated control tunnel.

DETAILED DESCRIPTION:
Background and aim:

Hidradenitis suppurativa (HS) is a common chronic skin disease that manifests by intermittent flare-ups of inflamed painful nodules that often leave mutilating scars, chronic suppurating tunnels and a changed microbiome compared to normal skin. Symptoms typically begin during adolescence and patients struggle with pain, pruritus, malodor and purulent discharge compromising work life, physical exercise, and sexual habits. Consequently, the risk of social exclusion, anxiety, depression and suicide is increased among patients suffering from HS.

Topical and systemic medical treatments, e.g. in the form of antibiotics, vitamin A derivates, immune-modulatory drugs or biological therapies aim to control inflammation. Once fistulas have formed, surgical intervention is often required. Present surgical therapies comprise surgical deroofing where the fistulas are cut open and left to heal, removal of specific pathological structures by ablative laser surgery or complete surgical removal en bloc of affected HS skin followed by skin grafting.

Recently, emergence of flexible diode laser fibers has enabled intra-lesional laser treatments of fistulas and the technique has been applied for e.g. perianal fistulas. Two prospective and one retrospective cohort studies evaluated a total of 265 patients treated with 1470 nm laser fiber surgery for perianal fistulas, demonstrating primary healing with absence of symptoms after one treatment in 40% to 71% of patients, a median healing time of 5 weeks, and long-term closure beyond 12 months in 71% of patients6. Intralesional laser fiber treatment has also been tested in HS tunnels. One study of concomitant 630 nm laser fiber treatment and photodynamic therapy has demonstrated a significant reduction in hidradenitis severity score and complete response in 47 % of patients after one treatment session.

Intralesional flexible laser fibers have also been tested in the treatment of HS tunnels without concomitant photodynamic therapy. One study investigated four sessions of 1064 nm intralesional diode laser therapy performed in local anesthesia. In a total of 20 patients, a significant reduction of Sartorius score and improved quality of life was demonstrated. No patients experienced neither worsening of disease nor complete cure and adverse effects were mild and transient. It was proposed, that intralesional laser treatment may elicit a decontaminating as well as an denaturing effect. Histological evaluation of endo-venous 1470 nm laser fiber treatment have demonstrated uniform coagulation without carbonization. Overall, the intralesional laser fiber technique is still new, and knowledge of optimal laser wave lengths, energy levels, number of treatments and treatment intervals is sparse. In addition, little is known about laser-tissue interactions in vivo as well as in vitro. However, there is reason to believe that intralesional laser fiber treatment of HS tunnels may provide a new tissue-sparing alternative to conventional surgical techniques with a potential to produce fewer side effects, less scaring, shorter downtime after surgery and possibly, also improved inflammatory control.

This study aims to investigate the efficacy and safety of 1470 nm laser fiber treatment of HS tunnels and add new knowledge of the microbiota as well as of laser-tissue interactions by in vivo ultrasound and in vitro histology.

Methods:

Study execution:

The project will be carried out at the Dermatological Department, Roskilde University Hospital under the leadership of principal investigator Professor Gregor Jemec, MD, DMSc. Senior doctor Ditte Marie Lindhardt Saunte, MD, PhD and Medical Doctor Elisabeth Hjardem Taudorf MD, PhD will run the project in cooperation with the established research group at the department

Study design:

A prospective cohort study of intralesional laser fiber treatment of HS fistulas is planned. Demographic data and information regarding prior treatments for HS will be collected in standardized case-report forms.

After signing informed consent, patients with HS tunnels in typical areas will be enrolled. Patients who have at least two suitable tunnels in typical HS areas will be invited to participate in the randomised within-person design to receive experimental laser fibre treatment. Two comparable HS tunnels from each patient will be selected enabling a subsequent randomisation to receive treatment or to serve as an intra-individual control, respectively.

Intervention:

The experimental treatment consists of one session of thermal coagulation with intralesional 1470 nm diode laser fibre in the entire length of one HS tunnel after injection of local anaesthetics (Mepivacaine-adrenaline). Both ends of tunnels selected for laser treatment must be accessible from the skin surface to ensure treatment of the entire tunnel.

ELIGIBILITY:
Inclusion Criteria:

* Legally competent women and men
* aged 18 years or older
* Two appropriate HS fistulas

Exclusion Criteria:

* fistulas in areas that have previously received surgery
* Allergy to lidocaine or adrenaline
* Fragile physical health that cannot tolerate standard of care HS rescue therapy
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
VAS pain | At baseline, 2, 6, and 12 weeks from baseline
  change in pain score on a visual analogue scale (where 0 is no pain =better; 10 is maximum pain = worse) for each individual HS-tunnel

SECONDARY OUTCOMES:
ultrasound | At baseline, and 12 weeks from baseline
  percentage closure of fistulas measured by ultrasound
Blinded evaluation of improvement of left/right tunnel (yes/no) in clinical photographs | At baseline, 2, 6 and 12 weeks post treatment
  Change in appearance of sets of photographs (treatment and control site). A blinded evaluator will be asked to evaluate improvement (yes/no) for each side.
Lesion count | At baseline, 2, 6 and 12 weeks post treatment
  Number of inflamed nodules and tunnels in each region
Change in Patients global assessment (PtGA) | At baseline, 2, 6 and 12 weeks post treatment
  Patient's overall evaluation of disease activity on a visual analogue scale (VAS) where 0 is no disease activity (=better); 100 is maximum disease activity (=worse)
Change in Physician's global assessment (PGA) | At baseline, 2, 6 and 12 weeks post treatment
  Physician's overall evaluation of disease activity on a visual analogue scale (VAS) where 0 is no disease activity (=better); 100 is maximum disease activity (=worse)
Described number of flares | At baseline, 2, 6 and 12 weeks post treatment
  Patient's description of number of flares since last appointment
Number of treated and control tunnels acquiring rescue therapy | At baseline, 2, 6 and 12 weeks post treatment
  The patient's need for rescue-treatment with intralesional triamcinolone in each tunnel since last appointment
Suppuration | At baseline, 2, 6 and 12 weeks post treatment
  degree of suppuration measured on a 4-point numerical ranking scale (0= no suppuration, 1=mild suppuration, 2 = moderate suppuration, 3 = severe suppuration)

OTHER OUTCOMES:
Changes in Microbiome by investigation of skin biopsies | At baseline and 6 weeks from baseline
  investigation of changes in skin microbiome in skin biopsies which will lead to descriptive observations of alterations in observed bacteria, vira and fungi
Thermography | At baseline, 2, 6, and 12 weeks from baseline
  Inflammation in each of the two tunnels as reflected by Thermography
Dermatology Life Quality index (DLQI) questionnaire | baseline
  Investigation of quality of life in this group of patients by a standardised dermatological questionaire. The questions relates to a standardized score between 0 and 30, where 0 means that the quality of life is not affected (better) and 30 means that quality of life is completely affected (worse).
Patient satisfaction: VAS | At 12 weeks from baseline
  Overall satisfaction with treatment on an overall on a visual analogue scale (VAS) where 0 is no satisfaction with treatment (=worse); 10 is maximum satisfaction with treatment (=better)
Number of patient preferring the treatment tunnel over the control tunnel | At 12 weeks from baseline
  Registration of which side (treated or control) the patients prefer over the other
Descriptive histological appearance of HS-tunnels | At baseline and 6 weeks from baseline
  Descriptive histological appearance of HS-tunnels and if possible, detection of histological changes after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gregor BE Jemec, DmSc, Prof., Principal Investigator — Zealand University Hospital - Roskilde
Locations (1):
- zealand University Hospital Roskilde, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Saunte DML, Jemec GBE. Hidradenitis Suppurativa: Advances in Diagnosis and Treatment. JAMA. 2017 Nov 28;318(20):2019-2032. doi: 10.1001/jama.2017.16691. PMID 29183082
- [Background] Ring HC, Thorsen J, Saunte DM, Lilje B, Bay L, Riis PT, Larsen N, Andersen LO, Nielsen HV, Miller IM, Bjarnsholt T, Fuursted K, Jemec GB. The Follicular Skin Microbiome in Patients With Hidradenitis Suppurativa and Healthy Controls. JAMA Dermatol. 2017 Sep 1;153(9):897-905. doi: 10.1001/jamadermatol.2017.0904. PMID 28538949
- [Background] Thorlacius L, Cohen AD, Gislason GH, Jemec GBE, Egeberg A. Increased Suicide Risk in Patients with Hidradenitis Suppurativa. J Invest Dermatol. 2018 Jan;138(1):52-57. doi: 10.1016/j.jid.2017.09.008. Epub 2017 Sep 20. PMID 28942360
- [Background] Terzi MC, Agalar C, Habip S, Canda AE, Arslan NC, Obuz F. Closing Perianal Fistulas Using a Laser: Long-Term Results in 103 Patients. Dis Colon Rectum. 2018 May;61(5):599-603. doi: 10.1097/DCR.0000000000001038. PMID 29528908
- [Background] Wilhelm A, Fiebig A, Krawczak M. Five years of experience with the FiLaC laser for fistula-in-ano management: long-term follow-up from a single institution. Tech Coloproctol. 2017 Apr;21(4):269-276. doi: 10.1007/s10151-017-1599-7. Epub 2017 Mar 7. PMID 28271331
- [Background] Giamundo P, Esercizio L, Geraci M, Tibaldi L, Valente M. Fistula-tract Laser Closure (FiLaC): long-term results and new operative strategies. Tech Coloproctol. 2015 Aug;19(8):449-53. doi: 10.1007/s10151-015-1282-9. Epub 2015 Feb 28. PMID 25724967
- [Background] Suarez Valladares MJ, Eiris Salvado N, Rodriguez Prieto MA. Treatment of hidradenitis suppurativa with intralesional photodynamic therapy with 5-aminolevulinic acid and 630nm laser beam. J Dermatol Sci. 2017 Mar;85(3):241-246. doi: 10.1016/j.jdermsci.2016.12.014. Epub 2016 Dec 19. PMID 28034606
- [Background] Fabbrocini G, Franca K, Lotti T, Marasca C, Annunziata MC, Cacciapuoti S, Masara A, Romanelli M, Lotti J, Wollina U, Tchernev G, Zerbinati N. Intralesional Diode Laser 1064 nm for the Treatment of Hidradenitis Suppurativa: A Report of Twenty Patients. Open Access Maced J Med Sci. 2018 Jan 7;6(1):31-34. doi: 10.3889/oamjms.2018.045. eCollection 2018 Jan 25. PMID 29483975